CLINICAL TRIAL: NCT00592735
Title: The Role of Adipocyte-derived Inflammatory Cytokines in the Pathogenesis of Diabetes, Dyslipidaemia, Atherosclerosis and Gastro-oesophageal Reflux Disease: the Effects of Medical and Surgical Weight Loss
Brief Title: Effects of Medical and Surgical Weight Loss on Metabolism
Acronym: BOS
Status: Completed | Type: Observational
Sponsor: Garvan Institute of Medical Research (Other)
Responsible Party: Principal Investigator, Professor Katherine Samaras, Professor Katherine Samaras, Garvan Institute of Medical Research
Other Study IDs: SVH H06/151; SVH H06/151
Record Dates: First submitted 2008-01-01; First posted 2008-01-14 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-06

CONDITIONS: Type 2 Diabetes; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Procedure: laparoscopic gastric banding

INTERVENTIONS:
Procedure: laparoscopic gastric banding — standard surgical procedure

SUMMARY:
This study will follow ,morbidly obese subjects as they undertake weight loss before and after laparoscopic gastric banding, examining markers of glucose and lipid metabolism, adipokines and measures of body fat.

ELIGIBILITY:
Inclusion Criteria:

* morbidly obese subjects with type 2 diabetes or metabolic syndrome
* age <70

Exclusion Criteria:

* contra-indications to bariatric surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: morbidly obese subjects with type 2 diabetes or metabolic syndrome
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2007-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
weight loss | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- St Vincent's Hospital, Sydney, New South Wales, Australia